CLINICAL TRIAL: NCT04323904
Title: Hantavirus Registry Gathers Knowledge on Epidemiology, Clinical Course, Prognostic Factors and Molecular Characteristics for Hantavirus Infections and Their Complications (HantaReg)
Brief Title: Hantavirus Registry - HantaReg
Acronym: HantaReg
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Principal Investigator, University of Cologne
Other Study IDs: HantaReg
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hantavirus Infections; Hemorrhagic Fever With Renal Syndrome; Nephropathia Epidemica; Hantavirus Cardiopulmonary Syndrome
MeSH Terms: conditions — Hantavirus Infections; Hemorrhagic Fever with Renal Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hantavirus Group: Patients with cultural, serological, molecular evidence of hantavirus infection
  Interventions: Other: Retrospective data collection
- Control group: Controls will be included at the same hospitals that conduced cases based on matching of demographics, underlying diseases and duration of hospitalization (i.e. one control per case, both in the same hospital)
  Interventions: Other: Retrospective data collection

INTERVENTIONS:
Other: Retrospective data collection — Retrospective data collection from patients with hantavirus infection and matching control group patients.

SUMMARY:
Hantavirus disease are zoonotic infections and remain a clinical challenge with globally increasing incidence and multiple serious outbreak situations in Europe within the last years. Hantavirus disease encompasses two clinical syndromes, hemorrhagic fever with renal syndrome (HFRS) and hantavirus cardiopulmonary syndrome (HCPS) caused by Old World and New World hantaviruses, respectively. Depending on the causative Old World hantavirus species, clinical course of HFRS can vary from mild to moderate to severe.

At present, there is no specific therapy available for hantavirus disease. As the clinical course of hantavirus disease is dependent on the causing viral pathogen and as there worrisome hints that clinical course HFRS and HCPS overlap, further studies with regard to the disease course are mandatory. Furthermore, the examination of attributable mortality and costs of hantavirus disease will need to be studied on a multinational basis and therefore HantaReg will particularly use a matched case control design.

DETAILED DESCRIPTION:
Hantavirus disease are zoonotic infections and remain a clinical challenge with globally increasing incidence and multiple serious outbreak situations in Europe within the last years. Hantavirus disease encompasses two clinical syndromes, hemorrhagic fever with renal syndrome (HFRS) and hantavirus cardiopulmonary syndrome (HCPS) caused by Old World and New World hantaviruses, respectively. Depending on the causative Old World hantavirus species, clinical course of HFRS can vary from mild to moderate to severe. HRFS caused by Hantaan virus, Amur virus and Dobrava-Belgrade virus lead to severe clinical course of the disease, with mortality ranging from 10-15%, whereas Seoul virus and Puumula virus result in mild to moderate from of disease with a mortality below <1%, also referred to as nephropathia epidemica. New World hantaviruses cause HCPS leading to acute respiratory distress syndrome (ARDS) and heart rhythm disorders with attributable mortality ranging high from 30-50%. However, there are hints that HRFS and HCPS overlap with a combined clinical course with cardiopulmonary, renal and hemorrhagic symptoms being present simultaneously. Due to climate changes and globalization, outbreak situations of hantavirus disease throughout Europe are increasing and there are worrisome trends regarding changing of species distributions in Europe.

At present, there is no specific therapy available for hantavirus disease. Treatment approaches are primarily supportive with admission of patients to the intensive care unit (ICU) and maintenance of fluid and electrolyte balance. Patients with severe renal insufficiency and fluid retention, pulmonary edema or hyperkalemia may require dialysis. In case of extensive thrombocytopenia and present bleeding, platelet transfusion may be needed. In HCPS, treatment approaches consist of the supplementation of oxygen, mechanical ventilation and in case of extended acute respiratory distress syndrome (ARDS) extracorporeal membrane oxygenation (ECMO).

Due to increasingly frequent outbreak situations and globally chances in species distributions, a worldwide surveillance in epidemiology and species attribution is needed. As the clinical course of hantavirus disease is dependent on the causing viral pathogen and as there worrisome hints that clinical course HFRS and HCPS overlap, further studies with regard to the disease course are mandatory. Furthermore, the examination of attributable mortality and costs of hantavirus disease will need to be studied on a multinational basis and therefore HantaReg will particularly use a matched case control design.

The objective of the Hantavirus Registry - HantaReg is to overcome the lack of knowledge on epidemiology, clinical course and prognostic factors for hantavirus infections and their complications, as well as to serve as a platform for future studies and outbreak situations.

ELIGIBILITY:
Inclusion Criteria:

* Serological or molecular evidence of hantavirus infection and clinical evidence of nephropathia epidemica or hemorrhagic fever with renal syndrome (HFRS)
* Serological or molecular evidence of hantavirus infection and clinical evidence of hantavirus cardiopulmonary syndrome (HCPS)

Exclusion Criteria:

- Serological or molecular evidence of hantavirus infection without clinical signs of nephropathia epidemica, HFRS or HCPS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with serological or molecular evidence of hantavirus infection and clinical evidence of nephropathia epidemica or hemorrhagic fever with renal syndrome (HFRS), or serological or molecular evidence of hantavirus infection and clinical evidence of hantavirus cardiopulmonary syndrome (HCPS).
  Particularly, controls will be identified retrospectively at the same hospitals that based on matching of demographics, underlying diseases and duration of hospitalization (i.e. one control per case, both in the same hospital).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence | up to 100 weeks
  To describe the global incidence of hantavirus infections
Mortality | up to 100 weeks
  To describe the global mortality due to hantavirus infections

SECONDARY OUTCOMES:
Complications | at 90 days from diagnosis
  To describe complications of hantavirus infections
Therapeutic approaches | at 90 days from diagnosis
  To describe therapeutic approaches of hantavirus infections
First-line and salvage treatment approaches | at 90 days from diagnosis
  To describe first-line and salvage treatment approaches and their efficacy and impact on patients' outcome
Recommendations for diagnosis and treatment | at 90 days from diagnosis
  To develop clinical screening and diagnostic approaches

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North-Rhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related information — http://www.kidneyinfection.org/leptoscope/